CLINICAL TRIAL: NCT06984250
Title: Hybrid Techniques Combining Hypofractionated Whole Breast Radiotherapy With Concomitant Tumor Bed Boost in Patients With Breast Cancer
Brief Title: Hypofractionated Radiotherapy With Concomitant Tumor Bed Boost for Breast Cancer
Acronym: HFCBB
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202110027RINB; 113-S0087 (Other Grant/Funding Number: National Taiwan University Hospital Yunlin Branch)
Record Dates: First submitted 2025-04-30; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-04

CONDITIONS: Early Breast Cancer; Ductal Breast Carcinoma In Situ
Keywords: breast cancer; concomitant boost; tumor bed; Intensity-modulated radiation therapy; hypofractionated breast radiotherapy
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- CBB: Hypofractionated breast radiotherapy following partial mastectomy in patients with early breast cancer or ductal breast carcinoma in situ
  Interventions: Radiation: Hypofractionated Radiation Therapy

INTERVENTIONS:
Radiation: Hypofractionated Radiation Therapy — Hypofractionated breast radiotherapy (HFRT) with hybrid techniques combining field-in-field intensity-modulated RT (FIF-IMRT) to the whole breast with inverse-IMRT for concomitant boost
  Other Names: Hypofractionated breast radiotherapy with concomitant boost

SUMMARY:
Hypofractionated breast radiotherapy with concomitant tumor bed boost for early breast cancer or ductal breast carcinoma in situ after partial mastectomy

ELIGIBILITY:
Inclusion Criteria:

* Female patients with histologically confirmed early-stage breast cancer (T1-2 and N0-1) or ductal carcinoma in situ (DCIS).
* Patients undergoing breast-conserving surgery
* Age ≥ 20 years
* Karnofsky Performance Status (KPS) ≥70%
* Life expectancy ≥ 5 years
* Adequate renal and hepatic function

Exclusion Criteria:

* Pregnant patients
* Patients requiring re-irradiation of the thoracic region

Ages: 20 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients diagnosed with early-stage breast cancer (T1-2 and N0-1) or ductal carcinoma in situ (DCIS) who are undergoing breast-conserving surgery.
Sampling Method: Probability Sample
Enrollment: 315 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2030-02-28 (Estimated)

PRIMARY OUTCOMES:
Ipsilateral breast tumor recurrence | From enrollment to the end of treatment at 2 years
  The time from the date of completion of radiotherapy to the date of ipsilateral breast recurrence or death, whichever occurs first. Unit of Measure: Time-to-event (months)

SECONDARY OUTCOMES:
Early Phase Acute Skin Toxicity | Up to 3 months following completion of radiotherapy
  Acute skin toxicity assessed using the Common Terminology Criteria for Adverse Events (CTCAE v5.0), grading severity from Grade 0 (none) to Grade 5 (death). Unit of Measure: CTCAE Grade (0-5)
Late Phase Breast Fibrosis | From 3 months up to 5 years following completion of radiotherapy
  Late breast fibrosis assessed using the Common Terminology Criteria for Adverse Events (CTCAE v5.0), grading severity from Grade 0 (none) to Grade 5 (death). Unit of Measure: CTCAE Grade (0-5)
Patient Quality of Life (EORTC QLQ-C30) | At baseline (before radiotherapy), between 1 week and 1 month following radiotherapy completion, then every 3 to 4 months thereafter until study completion (up to 5 years)
  Quality of life evaluation using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30), Chinese Mandarin (Taiwan) version. Scores range from 0 to 100, with higher scores indicating better quality of life. Unit of Measure: Score (0-100)
Patient Quality of Life (EORTC QLQ-BR23) | At baseline (before radiotherapy), between 1 week and 1 month following radiotherapy completion, then every 3 to 4 months thereafter until study completion (up to 5 years)
  Quality of life evaluation using the Breast Cancer Module (BR23) of the European Organization for Research and Treatment of Cancer, Chinese Mandarin (Taiwan) version. Scores range from 0 to 100, with higher scores indicating better quality of life. Unit of Measure: Score (0-100)

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Taipei, Taiwan
  - National Taiwan University Hospital Yunlin Branch, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Anonymized patient-level clinical data necessary to replicate the main study findings
Supporting Information: Study Protocol, SAP, CSR